CLINICAL TRIAL: NCT02229357
Title: Evaluation of Priming Effects by Pandemic Live Attenuated Influenza Vaccine (LAIV Candidate Vaccine Strain A/17/Turkey/Turkey/05/133 (H5N2)) on the Subsequent Response to Inactivated H5N1 Vaccine in Healthy Thai Volunteers: A Non-Randomized, Open Label Study
Brief Title: Evaluation of Priming Effects by PLAI Vaccine on the Subsequent Response to Inactivated H5N1 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government); World Health Organization (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GPO Avian Flu Vaccine-Boost
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Avian Influenza
Keywords: H5N2 Vaccine
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OrniFlu® inactivated vaccine (Experimental)
  Interventions: Biological: OrniFlu® inactivated vaccine

INTERVENTIONS:
Biological: OrniFlu® inactivated vaccine — All subjects will receive a single dose of an H5 inactivated influenza vaccine after blood collection for immunology assays

SUMMARY:
This study aim to compare immunogenicity of the inactivated H5 influenza vaccine single dose between subjects previously vaccinated with LAIV H5N2 and naïve subjects

DETAILED DESCRIPTION:
It is a non-randomized, open label study to evaluate a licensed OrniFlu® inactivated vaccine (produced by Microgen Russia) which will be given to healthy adult volunteers who participated in a double blind placebo-controlled study Protocol No.: GPO AVIAN FLU Vaccine-V02-2 at Vaccine Trial Centre and Department of Clinical Tropical Medicine, Faculty of Tropical Medicine, Mahidol University in February to May 2013.

A total of 60 subjects, of whom 40 received two doses of LAIV H5N2 (prime-boost group), and 20 received placebo (control group) in the previous study will be asked to return to the clinic to receive a single dose of an inactivated H5 influenza vaccine.

Total foloww up is 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Phase II study Protocol No.: GPO AVIAN FLU Vaccine-V02-2
* Healthy
* Age 18-49 years old
* Having Thai ID card or equivalent
* Anti HIV - Negative
* All hematology, biochemistry and urine analysis are within normal range or of no clinical significance (not higher than 1.5 time of normal value without any clinical finding from history and physical examination)
* Able to read and write and sign written informed consent.

Exclusion Criteria:

* Known history of egg allergy
* Having had recently influenza infection confirmed as H5
* Receiving other vaccination against H5N1
* History of bronchial asthma
* History of chronic lung diseases
* History of chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression< 6 months prior to immunization
* History of heavy smoking (more than 5 packs per day)
* History of alcoholic (pure drink 200 ml per day)
* Acute infectious and noninfectious diseases (within 2 weeks)
* HIV positives
* The volunteers who have been taking immunoglobulin products or have had a blood transfusion during past three months before the beginning of the experiment
* Participation in other research study or stop participant less than 1 month
* Pregnancy or plan to become pregnant for 60 days after enrollment or breast feeding
* Poultry workers

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects exhibiting sero-responses in each of the assays (HAI, microneutralization) in the prime-boost and the control groups. | 12 Months

SECONDARY OUTCOMES:
Post-vaccination injection site and systemic reactogenicity and adverse events to the H5 inactivated influenza vaccine in subjects previously primed with LAIV H5N2 and in naïve subjects. | 12 Month

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Principal Investigator — Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Pitisuttithum P, Boonnak K, Chamnanchanunt S, Puthavathana P, Luvira V, Lerdsamran H, Kaewkungwal J, Lawpoolsri S, Thanachartwet V, Silachamroon U, Masamae W, Schuetz A, Wirachwong P, Thirapakpoomanunt S, Rudenko L, Sparrow E, Friede M, Kieny MP. Safety and immunogenicity of a live attenuated influenza H5 candidate vaccine strain A/17/turkey/Turkey/05/133 H5N2 and its priming effects for potential pre-pandemic use: a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2017 Aug;17(8):833-842. doi: 10.1016/S1473-3099(17)30240-2. Epub 2017 May 19. PMID 28533093